CLINICAL TRIAL: NCT05569239
Title: Phase 2b, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Immunogenicity and Safety of One Dose of OVX836 Influenza Vaccine 480μg, After Intramuscular Administration in Healthy Subjects Aged 18-59 Years
Brief Title: Efficacy, Immunogenicity and Safety of OVX836 Influenza Vaccine 480μg
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Osivax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OVX836-005
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: A total number of 2,850 subjects are planned to be randomized (in a 1:1 ratio) into 2 groups to receive a single intramuscular injection of either OVX836 (480μg) or placebo.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OVX836 480µg (Experimental): Adjuvant-free recombinant influenza candidate vaccine based on Nucleoprotein in the influenza virus. One single administration intramuscularly of 480µg dose on Day1.
  Interventions: Biological: OVX836 480µg
- Placebo (Placebo Comparator): Saline solution (B. Braun Ecoflac Plus) Saline solution (Nacl 0.9%), B. Braun Ecoflac Plus 50mL. One single administration intramuscularly of a 0.8mL dose on Day1.
  Interventions: Biological: Saline Solution

INTERVENTIONS:
Biological: OVX836 480µg — One single administration intramuscularly at Day 1.
  Arms: OVX836 480µg
Biological: Saline Solution — One single administration intramuscularly at Day 1.
  Arms: Placebo

SUMMARY:
The present study will evaluate the efficacy, immunogenicity and safety of one dose of OVX836 influenza vaccine 480μg, after intramuscular administration in healthy subjects aged 18-59 years.

DETAILED DESCRIPTION:
This Phase 2b proof-of-concept field efficacy study is designed as a randomized, double-blind, parallel groups, placebo-controlled, multi-country, multicenter clinical trial. This design of prospective interventional trial is the gold standard in evaluating absolute efficacy of a product in preventing a disease or an outcome. An adequate number of observations is ensured by the multicenter approach.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Healthy male or female subjects, as determined by medical history and medical examination.
3. Between the ages of 18 and 59 years, inclusive.
4. Subject socially active: living in a family with children or with other house-hold members, having frequent social contacts at university, work, in public places such as restaurants, theaters, public transportation, etc.
5. Subjects compliant with the reproductive criteria for male and female participants .
6. Reliable and willing to make themselves available for the duration of the study, and willing and able to follow study procedures
7. Able to read, understand and complete an electronic Diary and electronic Patient Reported Outcome.
8. Able to read and sign the subject information sheet and informed consent form (ICF).

Exclusion Criteria:

1. Previous vaccination with an authorized or experimental seasonal, zoonotic or pandemic influenza vaccine within 6 months before the day of vaccination or planned to receive it during the whole study period.
2. Formal indication for influenza vaccination on an individual basis according to local recommendations, for example based on occupational risk, or underlying medical conditions. An informed subject who would refuse to get the regular influenza vaccination would be allowed to participate in this study.
3. Any known or suspected immunodeficient conditions.
4. Past or current history of significant autoimmune diseases, as judged by the Investigator.
5. Known or suspected infection with human immunodeficiency virus, hepatitis C virus, or hepatitis B virus.
6. Current history of significant uncontrolled medical illness such as diabetes, hypertension, heart, renal or hepatic diseases, as judged by the Investigator.
7. Planned absences without access to the investigational site, i.e. vacation or business trips, for more than 7 consecutive days during the study period
8. Pregnant or lactating woman.
9. Females planning to become pregnant or planning to discontinue contraceptive precautions until the end of the trial.
10. Having received another vaccine within 1 month prior to the day of study vaccination, except COVID-19 vaccines for which the minimum time period should be two weeks prior to study vaccination.
11. Having participated or currently participating in an OVX836 study or in the OVX-FLU-002 study.
12. Planning to receive any other vaccines during the first 28 days following the study vaccine administration, except COVID-19 vaccines which can be administered from 14 days following the study vaccine administration.
13. Administration of any investigational or non-registered drug or vaccine within 1 months prior to the administration of study vaccines, or planned administration of any such product during the whole study period.
14. History of receiving blood, blood components or immunoglobulins within 3 months prior to the day of vaccination, or planned to receive such product during the whole study period.
15. Presence of an acute febrile illness on the day of planned vaccination (oral temperature >38.0°C; temporary exclusion criterion).

16Diagnosed long COVID-19 subjects. 17. Presence of a condition in the ear-nose-throat area, such as nasal septum deviation, atrophic rhinitis, etc…, that could render nasal and nasopharyngeal swabs more difficult to perform, or increase the risk of bleeding; to be confirmed by medical history question and inspection of nasal passage.

18. Past or current history of any progressive or severe uncontrolled neurological disorder, seizure disorder or Guillain-Barré syndrome.

19. Behavioral or cognitive impairment, or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the study.

20. Past (stopped less than 6 months before enrolment) or current smoking habit above 10 cigarettes per day.

21. Past (stopped less than 6 months before enrolment) or current history of heavy alcohol use, defined as follows: for men, consumption of more than 4 standard drinks on any day or more than 14 standard drinks per week, and for women, consumption of more than 3 standard drinks on any day or more than 7 standard drinks per week.

22. Past (stopped less than 6 months before enrolment) or current use of recreational drugs, which could interfere with the adherence to the protocol procedures.

23. Chronic or prolonged treatment (>10 consecutive days) that can affect immune response, such as systemic (≥ 20 mg/day prednisone or equivalent or dexamethasone >4 mg/day), high dose inhaled corticosteroids (>800 μg/day beclomethasone or equivalent; occasional inhaled, topical or localized injections [intra-articular or intra-bursal] of corticosteroids for asthma therapy are allowed), or immunomodulators/suppressors (certain monoclonal antibodies can be approved on a case by case basis) within 28 days before study entry or during the whole study duration.

24. Chronic or prolonged (>10 days) use of systemic non-steroidal anti-inflammatory drugs, acetylsalicylic acid, or paracetamol within 7 days before study entry and up to 28 days post-vaccination.

25. Prophylactic or therapeutic use of influenza antivirals within 7 days prior to the day of study vaccination or during the whole study duration.

26. History of severe allergic reactions and/or anaphylaxis, or serious adverse reactions to vaccines or allergy to kanamycin or any other component of the OVX836 vaccine.

27. Any contraindication to intramuscular administration, as judged by the Investigator.

28. Presence of extended tattoos on both deltoid muscles. 29. Individuals with history of any illness that, in the opinion of the Investigator, might interfere with the results of the study, or pose additional risk to the subjects due to participation in the study, either directly or through any treatments administered for that illness.

30. Sponsor employees or Investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse (or assimilated), parent, child or sibling, whether biological or legally adopted.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2850 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
First occurrence of RT-PCR-confirmed influenza Type A symptomatic disease | During the whole study duration, up to maximum 10 months

SECONDARY OUTCOMES:
First occurrence of RT-PCR-confirmed influenza symptomatic disease irrespective of strain/type. | During the whole study duration, up to maximum 10 months.
First of occurrence of RT-PCR-confirmed influenza Type B symptomatic disease | During the whole study duration, up to maximum 10 months
Number of subtype of virus in RT-PCR-confirmed influenza Type A cases. | During the whole study duration, up to maximum 10 months
Severity and duration of Influenza Like Illness episodes | During the whole study duration, up to maximum 10 months
First occurence of clinical influenza-like disease irrespective of causal agent | During the whole study duration, up to maximum 10 months
Number of occurence of solicited local and systemic signs and symptoms | During 7 days after vaccine administration
Number of occurence of subjects reporting unsolicited AEs | During 29 days after vaccine administration
Number of occurence of subjects reporting Serious Adverse Events, Adverse Events of Special Interest, New Onset of Chronic Disease, Medical Attended Adverse Events | During the whole study period, maximum 10 months
Cell-mediated immune response in Peripheral Blood Mononuclear Cells, measured by Interferon Gamma Enzyme-Linked Immunospot Assay in a limited subset of 56 subjects. | At Day 1 and Day 8
  Elispot
Number and percentage of subjects with NP-specific T-cell measured by Interferon Gamma Enzyme-Linked Immunospot Assay. | At Day 1 and Day 8
  Elispot
Percentage of NP specific CD4+ and CD8+ T-cell measured by flow cytometry on PBMCs as expressing IL-2, TNFα and/or IFNγ at pre-injection baseline (Day 1) | At Day 1 and Day 8
  ICS
Number and percentage of subjects with a percentage of NP specific CD4+ and CD8+ T-cell expressing IL-2, TNFα and/or IFNγ at Day 8 or Day 29 higher than the percentile 95 of the pre-injection baseline (Day 1) | At Day 1 and Day 8
  ICS
Geometric Mean Titer of anti-Nucleoprotein immunoglobulin G (Enzyme-Linked Immunosorbent Assay, serum). | At Day 1 and Day 8
  Elisa
Number and percentage of subjects with a four-fold increase of anti-Nucleoprotein immunoglobulin G (Enzyme-Linked Immunosorbent Assay, serum) titre with respect to pre-injection baseline (Day 1) | At Day 1 and Day 8
  Elisa
Percentage of NP specific CD4+ and CD8+ T-cell measured by flow cytometry on PBMCs as expressing IL-2, TNFα and/or IFNγ in a limited subset of 56 subjects | At Day 1 and Day 8
  ICS
Anti-Nucleoprotein immunoglobulin G measured by Enzyme-Linked Immunosorbent Assay in, serum in a limited subset of 56 subjects. | At Day 1 and Day 8
  Elisa

CONTACTS AND LOCATIONS:
Locations (16):
- Belgium (4):
  - Site BE-02, Antwerp
  - Site BE-03, Antwerp
  - Site BE-01, Ghent
  - Site BE-04, Mechelen
- Finland (8):
  - Site FI-12, Espoo
  - Site FI-08, Helsinki
  - Site FI-13, Jarvenpaa
  - FI-14, Kokkola
  - Site FI-11, Oulu
  - Site FI-15, Seinäjoki
  - Site FI-09, Tampere
  - Site FI-10, Turku
- France (3):
  - Site FR-05, Lyon
  - Site FR-07, Paris
  - Site FR-06, Rennes
- Site DE-16, München, Germany

IPD SHARING:
Plan to Share IPD: No